CLINICAL TRIAL: NCT06996535
Title: Pancreatic Quantitative Sensory Testing (P-QST) in Pediatric Patients With Acute Recurrent Pancreatitis and Chronic Pancreatitis: Evaluation and Prediction of Treatment Response
Brief Title: Pancreatic Quantitative Sensory Testing (P-QST)
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0046
Record Dates: First submitted 2023-11-27; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pancreatitis; Chronic Pain; Acute Recurrent Pancreatitis
Keywords: Pediatric
MeSH Terms: conditions — Pancreatitis, Chronic; Chronic Pain | interventions — Postsynaptic Potential Summation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Controls: Subjects with no pancreatic disease and no abdominal pain.
  Subjects will undergo the following Interventions:
  Quantitative Sensory Test 1, Quantitative Sensory Test 2, and Quantitative Sensory Test 3, They will also fill out validated questionnaires.
  Interventions: Diagnostic Test: Quantitative Sensory Test 1; Diagnostic Test: Quantitative Sensory Test 2; Diagnostic Test: Quantitative Sensory Test 3
- Chronic Pancreatitis patients: Quantitative Sensory Test 1, Quantitative Sensory Test 2, and Quantitative Sensory Test 3, They will also fill out validated questionnaires.
  Interventions: Diagnostic Test: Quantitative Sensory Test 1; Diagnostic Test: Quantitative Sensory Test 2; Diagnostic Test: Quantitative Sensory Test 3

INTERVENTIONS:
Diagnostic Test: Quantitative Sensory Test 1 — Subject will give pain rating (on Visual Analogue Scale (VAS) 0-10) of single as well as multiple stimulation with round-tip non-invasive pin-prick device. Difference is recorded as Temporal Summation Score.
  Other Names: Temporal Summation
Diagnostic Test: Quantitative Sensory Test 2 — Subject will state when they first detect pain and pain detection threshold in response to pressure administration with pressure algometer. Pressure threshold recorded in kilopascals(kP). Stimulation will be repeated in pancreatic and control dermatomes. Subject will then state pain tolerance threshold at same locations. Sensitization will be characterized by ratio of pancreatic vs. control dermatome scores.
  Other Names: Segmental v Systemic Sensitization
Diagnostic Test: Quantitative Sensory Test 3 — Subject will apply dominant hand to ice-chilled water bath (36F) for up to 2 minutes. Pain score (VAS 0-10) will be assessed each 10 seconds. Pain tolerance threshold (in kP) will be assessed with algometer on non-dominant thigh before and after water bath to determine change in threshold. Difference in pain tolerance recorded as Conditioned Pain Modulation Score.
  Other Names: Conditioned Pain Modulation

SUMMARY:
Quantitative Sensory Testing (QST) is a novel investigative technique used in other pain conditions to evaluate patterns of chronic pain, and in this study will be used to elucidate pain patterns in patients with Chronic Pancreatitis (CP). QST uses a specific series of standardized stimulations to map the pain system. QST has the potential to change and improve the treatment paradigm for patients with CP and may eventually be able to predict response to invasive CP therapies.

DETAILED DESCRIPTION:
In Chronic Pancreatitis (CP), clinical pain symptoms correlate poorly with pancreatic ductal morphology, response to endoscopic or surgical therapy is unpredictable, and the rationale for invasive therapies is often questioned. Quantitative sensory testing (QST) is a technique used to map the pain system based on the rationale that different neural pathways and networks can be explored using standardized stimulation and simultaneous recording of the evoked pain response by psychophysical and/or objective methods. In this study, the investigators aim to distinguish phenotypes characterized by segmental sensitization of the pancreatic viscerotome, and systemic sensitization with pathological central pain processing.

The investigators will perform QST on controls and CP subjects consisting of stimulation in several different dermatomes including pancreatic and control areas. All subjects will also answer standardized questionnaires assessing pain, depression, anxiety, and quality of life at baseline. Subjects undergoing endoscopic or surgical therapy will also undergo follow-up testing consisting of the same tests at 3, 6, and 12 months post-procedure for evaluation of changes in their pain profile.

ELIGIBILITY:
Subjects with no pancreatic disease and no abdominal pain.

Inclusion Criteria:

* Subjects are 5 years to 17 years old
* Subject and or legal guardian is willing and able to comply with the scheduled visits, questionnaires, treatment plan, and other study procedures.
* Subjects with evidence or history of medical or surgical disease of importance for this study as judged by investigator.
* Subjects suffering from painful conditions that make them unable to distinguish the pain associated with ARP or CP from chronic pain of other origins.

Exclusion Criteria:

* • Subjects with evidence or history of medical or surgical disease of importance for this study as judged by investigator.

  * Subjects suffering from painful conditions that make them unable to distinguish the pain associated with ARP or CP from chronic pain of other origins.

Definite Chronic Pancreatitis

Inclusion Criteria: • Subjects are 5 years to 17 years old

* Subjects will have a prior confirmed diagnosis of CP on CT scan or MRI/MRCP according to Cambridge Classification (grade 3 or 4)
* Subjects and or legal guardian willing and able to comply with the scheduled visits, questionnaires, and other study procedures.

Exclusion Criteria:

* Subjects with evidence or history of medical or surgical disease of importance for this study as judged by investigator.
* Subjects suffering from painful conditions other than pancreatitis or SOD type 1 or 2 that make them unable to distinguish the pain associated with pancreatitis or SOD from chronic pain of other origins.
* Subjects with known pregnancy at the time of enrollment.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Stratified Sampling
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain Pattern Assessment | day 1
  Pain Pattern Assessment as assessed by the combination of Temporal Summation score, Sensitization score, and Conditioned Pain Modulation score

CONTACTS AND LOCATIONS:
Overall Officials: Juan Gurria, Principal Investigator — Cincinnati Childrens Hospital Medical Center
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No